CLINICAL TRIAL: NCT00238615
Title: A Phase II Trial of Concurrent Docetaxel (Taxotere) / Carboplatin / Radiotherapy Followed by Surgical Resection Followed by Consolidation Taxotere / Carboplatin in Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase II Docetaxel / Carboplatin / XRT + Surgical Resection in Stage III NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Stanford University (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Heather Wakelee, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN0002; 78999 (Other: Stanford University Alternate IRB Approval Number); GIA #12169 (Other: Aventis); 11804 (Other: Stanford IRB)
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Results first posted 2013-07-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Lung Cancer; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Carboplatin; Radiotherapy; Radiation; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy+Radiation+Surgery (Experimental): 1. Concurrent weekly docetaxel at 20 mg/m2 and weekly carboplatin at an AUC of 2 with thoracic radiotherapy of 180-200cGy/day for 5/7 days to 45 Gy.
  2. Complete surgical excision 3-6 weeks after completion of chemoradiotherapy.
  3. No Surgery if patient is deemed unable to tolerate surgery, with completion to 61 Gy radiation
  4. Consolidation after surgery: Docetaxel given at 75 mg/m2 every 3 weeks with carboplatin at AUC 6 every 3 weeks with concomitant growth factor support.
  Interventions: Drug: Docetaxel; Drug: Carboplatin; Procedure: Radiation therapy; Procedure: Surgical resection

INTERVENTIONS:
Drug: Docetaxel — 20 mg/m2, 75 mg/m2 infusion
  Other Names: Taxotere
Drug: Carboplatin — AUC of 2 and 6 infusion
  Other Names: Paraplatin
Procedure: Radiation therapy — NEOADJUVANT RADIOTHERAPY Radiation therapy will be concurrent with the chemotherapy. Radiation therapy will begin within 24 hours of chemotherapy. CONSOLIDATION RADIOTHERAPY Patients with positive surgical margins or incomplete resection (tumor shaved from spine or great vessels) will receive an additional boost of radiotherapy 3 to 6 weeks after surgery. This will be a 16 Gy boost given with concurrent weekly chemotherapy as during the neoadjuvant period.
  Other Names: radiation oncology; radiotherapy
Procedure: Surgical resection — All patients will be taken to surgical excision, unless they have developed a condition other than progressive disease, which would make surgery unsafe.
  Other Names: segmentectomy; segmental resection

SUMMARY:
The purpose of this study is to assess how well this particular combination of chemotherapy, radiation and surgery works to help people with locally advanced lung cancer, how well PET scans indicates whether someone has responded to chemotherapy and radiation, and gene expression patterns related to outcomes in patients with locally advanced lung cancer who receive this treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed stage IIIA or IIIB NSCLC

* Patients must have measurable disease
* No previous chemotherapy, radiation therapy or other systemic therapy for their NSCLC.
* Age>18 years
* Life expectancy >12 months
* ECOG performance status 0-1
* Normal organ and marrow function
* Medically fit for surgery at time of enrollment.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of the study. Women must have a negative pregnancy test prior to enrollment.
* Ability to understand and willingness to sign the consent form.

Exclusion Criteria:

* Previous chemotherapy, radiation therapy or any other systemic treatment for their NSCLC.
* Patients receiving any other investigational agents.
* Known metastatic disease (brain or any other site)
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 or with allergic reactions to compounds of similar chemical composition to carboplatin or other agents used in the study.
* Peripheral neuropathy >grade 1
* Uncontrolled concurrent illness
* Pregnant women
* Weight loss>10% in the past 3 months before diagnosis.
* Hyperglycemia - exclusion from PET analysis
* HIV positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with docetaxel and carboplatin or other agents administered during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2003-03; Primary Completion 2009-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather A. Wakelee, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Kozak MM, Murphy JD, Schipper ML, Donington JS, Zhou L, Whyte RI, Shrager JB, Hoang CD, Bazan J, Maxim PG, Graves EE, Diehn M, Hara WY, Quon A, Le QT, Wakelee HA, Loo BW Jr. Tumor volume as a potential imaging-based risk-stratification factor in trimodality therapy for locally advanced non-small cell lung cancer. J Thorac Oncol. 2011 May;6(5):920-6. doi: 10.1097/jto.0b013e31821517db. PMID 21774104
- [Result] Das M, Donington JS, Murphy J, Kozak M, Eclov N, Whyte RI, Hoang CD, Zhou L, Le QT, Loo BW, Wakelee H. Results from a single institution phase II trial of concurrent docetaxel/carboplatin/radiotherapy followed by surgical resection and consolidation docetaxel/carboplatin in stage III non-small-cell lung cancer. Clin Lung Cancer. 2011 Sep;12(5):280-5. doi: 10.1016/j.cllc.2011.06.003. Epub 2011 Jul 14. PMID 21752720

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel / Carboplatin / XRT + Surgical Resection: Patients were treated on this prospective phase II trial of trimodality therapy. Induction treatment consisted of weekly docetaxel 20 mg/m2 and weekly carboplatin at an area under curve (AUC) of 2 concurrent with 45 Gy thoracic radiotherapy. Resection was performed unless felt to be unsafe or if patients had progressive disease. Postoperative consolidation consisted of docetaxel 75 mg/m2 and carboplatin at an AUC of 6 every 3 weeks for 3 cycles with growth factor support. Patients were followed for survival outcomes.
Period: Overall Study
Arm/Group | Docetaxel / Carboplatin / XRT + Surgical Resection
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Secondary Outcome: Change in Standard Uptake Value (SUVmax) on Positron Emission Tomography (PET) Scans Pre and Post Chemotherapy and Radiation in This Trial and Ability to Predict Surgical Resection Rate, Progression-free Survival and 2 Year Overall Survival
Description: The change in standardized uptake values (SUV)max on PET scans obtained pre- and after 5 weeks of combined chemo-radiation for patients enrolled on the trial were evaluated for ability to predict outcomes including complete resection at time of surgery (3-6 weeks after completion of the chemo-radiation), progression-free survival and 2 year overall survival. The mean SUVmax pre chemoradiation minus the mean SUVmax post-radiation is reported.
Time Frame: baseline, 5 weeks after combined chemo-radiation
Population: All enrolled patients were analyzed in the published manuscript
Measure: Mean (Standard Deviation); unit: standardized uptake value (SUV)max
Groups:
- Docetaxel / Carboplatin / XRT + Surgical Resection: All patients enrolled had combined chemotherapy/radiation followed by surgical resection (other than 1 patient who had only chemotherapy/radiation) and were evaluated for a primary endpoint of 2 year overall survival. PET scans obtained pre and post 5 weeks of combined therapy were analyzed for predictive capacity relative to this endpoint.
  Results were published PMID 21774104
Arm/Group | Docetaxel / Carboplatin / XRT + Surgical Resection
Number analyzed (Participants) | 13
standardized uptake value (SUV)max | 5.7 (5.3)

2. Other Pre Specified Outcome: Exploratory Analysis of Relation of Gene Expression Patterns to Outcomes in Patients With Locally Advanced Lung Cancer Who Receive This Treatment Regimen
Description: This analysis of gene expression patterns related to outcomes in patients with locally advanced lung cancer who received this treatment regimen was not performed due to lack of funding.
Time Frame: Specimen collected at time of surgery
Population: Plan was to analyze all patients with adequate tissue for this analysis, but was not done. We did not have sufficient funds for this analysis.
Groups:
- Docetaxel / Carboplatin / XRT + Surgical Resection: This planned analysis of gene expression patterns was not performed.
Arm/Group | Docetaxel / Carboplatin / XRT + Surgical Resection
Number analyzed (Participants) | 0

3. Primary Outcome: 2 Year Overall Survival After a Combination of Chemotherapy, Radiation and Surgery in Stage III NSCLC Patients Following the Protocol Therapy.
Description: Patients were analyzed for 2 year overall survival after receiving trimodality (chemotherapy/radiation/surgery) therapy for stage III NSCLC. Patients had a chest x-ray and a doctor visit with a physical examination every 3 months after completion of all therapy for 3 years then every 6 months for 3 years to look for evidence of recurrent disease and to follow survival. Thoracic computed tomography (CT) scans were obtained at 6, 12, 18 months after completion of all therapy and then yearly for 3 years or as clinically indicated to evaluate for relapse.
Time Frame: Two years
Population: All patients alive and not censored at 2 years
Measure: Number; unit: participants
Groups:
- Docetaxel+Carboplatin +Radiation+Surgery: Patients were treated on this prospective phase II trial of trimodality therapy. Induction treatment consisted of weekly docetaxel 20 mg/m2 and weekly carboplatin at an area under curve (AUC) of 2 concurrent with 45 Gy thoracic radiotherapy. Resection was performed unless felt to be unsafe or if patients had progressive disease. Postoperative consolidation consisted of docetaxel 75 mg/m2 and carboplatin at an AUC of 6 every 3 weeks for 3 cycles with growth factor support. Patients were followed for survival and progression free survival outcomes.These results are published PMID: 21752720.
Arm/Group | Docetaxel+Carboplatin +Radiation+Surgery
Number analyzed (Participants) | 13
participants | 7
Statistical Analysis 1: Comparison: Docetaxel+Carboplatin +Radiation+Surgery; 2-year overall survival (OS) Our null hypothesis was a probability of survival at 2 years of 0.30. The study was powered at 80% (with α 5% two-tailed) to detect a probability of survival at 2 years of 0.55. This would require 30 patients assuming accrual over 2 years with 1 year of additional follow-up. The probability of survival at 2 years of 0.55 is based on previous studies of neoadjuvant approaches with reported 2 year survival in the 40-60% range; Test type: Superiority or Other; The primary endpoint of 2 year overall survival was (0.72) = 72%; probability of survival at 2 years = .72, 95% CI 2-sided [0.36 to 0.90], Standard Deviation 0

ADVERSE EVENTS:
Time Frame: Patients were followed for toxicity through completion of all protocol defined therapy (approximately 5 months) and for an additional month after completed of all therapy for toxicity (a total of 6-7 months).
Groups:
- Docetaxel / Carboplatin / XRT + Surgical Resection: Adverse events for all enrolled patients were followed. Details are published in PMID: 21752720
Arm/Group | Docetaxel / Carboplatin / XRT + Surgical Resection
Serious Adverse Events (participants affected / at risk) | 8/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel / Carboplatin / XRT + Surgical Resection (N=13)
esophagitis (Gastrointestinal disorders) | 1 (1) — 1 Grade III during indcution
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
anemia (Blood and lymphatic system disorders) | 2 (2)
neutropenia (Blood and lymphatic system disorders) | 1 (2)
allergic reaction (Injury, poisoning and procedural complications) | 2 (3)
fatigue (General disorders) | 4 (4)
dehydration (Metabolism and nutrition disorders) | 1 (1)
bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Resolved with conservative management (no surgical intervention required).
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Docetaxel / Carboplatin / XRT + Surgical Resection (N=13)
anemia (Blood and lymphatic system disorders) | 2 (4)
fatigue (General disorders) | 5 (5)
esophagitis (Gastrointestinal disorders) | 5 (5)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Accrual was very slow. The study was halted with accrual of only 13 patients. These results were published.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No